CLINICAL TRIAL: NCT07323407
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Transcranial Alternating Current Stimulation (tACS) for the Treatment of Refractory Constipation Comorbid With Somatic Symptom Disorder
Brief Title: Transcranial Alternating Current Stimulation for Refractory Constipation With Somatic Symptom Disorder
Acronym: RELIEF-tACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhifeng Zhao, PhD, Principal Investigator, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJLL-KY-20252521
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Functional Constipation (FC); Somatic Symptom Disorder (DSM-5); Refractory Constipation
Keywords: Functional Constipation; Somatic Symptom Disorder; refractory constipation; transcranial alternating current stimulation
MeSH Terms: conditions — Constipation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, placebo-controlled "Parallel Assignment" design with two arms:
  Experimental Arm - transcranial alternating current stimulation (tACS)
  Control Arm - Matching Placebo
  Participants are assigned in a 1 : 1 ratio by a central interactive web-response system, using permuted blocks stratified by study center and baseline CSBM frequency. Each participant receives only one intervention for the entire 4-week treatment period (plus taper/follow-up), with no crossover between arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tACS (Experimental): Electrode placement: Referenced to the forehead (Fpz) and bilateral mastoid regions, covering the prefrontal cortex and related brain-gut axis pathways.
  Stimulation parameters: Alternating current, 15 mA intensity, 77.5 Hz frequency.
  Dosing schedule: Once daily, 30-40 minutes per session, for 4 consecutive weeks (20 sessions total; Monday-Friday with weekend breaks).
  Interventions: Device: Transcranial Alternating Current Stimulation
- Placebo (Placebo Comparator): Electrode placement: Same as active-referenced to the forehead (Fpz) and bilateral mastoid regions, to mimic coverage of the prefrontal cortex and related brain-gut axis pathways.
  Stimulation parameters: Sham stimulation; the device is programmed to deliver a brief ramp-up and ramp-down at session start (e.g., ≤30 seconds total) to reproduce initial skin sensations, followed by no sustained current (0 mA effective intensity; no therapeutic stimulation).
  Dosing schedule: Once daily, 30-40 minutes per session, for 4 consecutive weeks (20 sessions total; Monday-Friday with weekend breaks).
  Blinding procedures: Device display, sounds, and electrode preparation identical to the active arm; session duration and operator interactions matched to maintain participant and assessor blinding.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Electrode placement: Referenced to the forehead (Fpz) and bilateral mastoid regions, covering the prefrontal cortex and related brain-gut axis pathways.
  Stimulation parameters: Alternating current, 15 mA intensity, 77.5 Hz frequency.
  Dosing schedule: Once daily, 30-40 minutes per session, for 4 consecutive weeks (20 sessions total; Monday-Friday with weekend breaks).
  Arms: tACS
Device: Placebo — Electrode placement: Same as active-referenced to the forehead (Fpz) and bilateral mastoid regions, to mimic coverage of the prefrontal cortex and related brain-gut axis pathways.
  Stimulation parameters: Sham stimulation; the device is programmed to deliver a brief ramp-up and ramp-down at session start (e.g., ≤30 seconds total) to reproduce initial skin sensations, followed by no sustained current (0 mA effective intensity; no therapeutic stimulation).
  Dosing schedule: Once daily, 30-40 minutes per session, for 4 consecutive weeks (20 sessions total; Monday-Friday with weekend breaks).
  Blinding procedures: Device display, sounds, and electrode preparation identical to the active arm; session duration and operator interactions matched to maintain participant and assessor blinding.
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled trial is to evaluate the efficacy and safety of transcranial alternating current stimulation (tACS) in adults with refractory functional constipation comorbid with somatic symptom disorder. This population is characterized by persistent bowel dysfunction despite conventional treatments, frequent reliance on laxatives, and evidence of impaired brain-gut regulation contributing to chronic symptoms.

The study focuses on three primary domains:

Efficacy - Bowel Function:

• Assessment of whether a 4-week course of tACS improves bowel activity, measured by changes in Complete Spontaneous Bowel Movements (CSBM) and overall bowel-movement frequency over the treatment and follow-up period.

Efficacy - Symptom and Quality of Life Burden:

• Evaluation of the effect of tACS on constipation-related severity and patient-reported outcomes, including the Patient Assessment of Constipation-Symptoms (PAC-SYM) and Patient Assessment of Constipation-Quality of Life (PAC-QOL).

Safety and Tolerability:

• Documentation of adverse events associated with tACS, with particular attention to incidence, intensity, and overall patient tolerability compared with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Functional Constipation (FC): Subjects must meet the diagnostic criteria for functional constipation as defined by the Rome IV criteria.
2. Low Frequency of Complete Spontaneous Bowel Movements (CSBM): During the 2-week screening period, subjects must have ≤2 complete spontaneous bowel movements per week.
3. Poor Response to Previous Treatment: Subjects must have been dissatisfied with prior treatments for functional constipation and have undergone at least 3 months of therapy (including laxatives or other prokinetic agents).
4. Diagnosis of Somatic Symptom Disorder (SSD): Subjects must meet the DSM-5 diagnostic criteria for somatic symptom disorder (SSD). All subjects will undergo a semi-structured clinical interview based on DSM-5 criteria, conducted by professionals trained in SSD diagnosis.

   * Criterion A: Presence of one or more distressing somatic symptoms that significantly affect daily life.
   * Criterion B: At least one of the following must be met:

     1. Excessive and persistent thoughts about the severity of symptoms;
     2. Persistently high levels of anxiety about health or symptoms;
     3. Excessive time and energy devoted to health concerns or symptoms.
   * Criterion C: Symptoms must persist for at least 6 months.
5. Age Range: Subjects must be between 18 and 80 years old.
6. No Concurrent Clinical Trials: Subjects must not participate in any other clinical trials during the study period.
7. Informed Consent: Subjects must voluntarily agree to participate and sign an informed consent form.

Exclusion Criteria:

1. Presence of organic diseases (such as tuberculosis, polyps, Crohn's disease, tumors, congenital megacolon, etc.), endocrine disorders (e.g., hypothyroidism), metabolic diseases (diabetes, thyroid dysfunction), or neurological disorders (e.g., Parkinson's disease);
2. Long-term use of medications that may affect intestinal function or induce constipation, such as Parkinson's drugs (excluding conventional laxatives, antidiarrheals, or intestinal stimulants; during the trial, participants are only allowed to take prescribed emergency medications, with detailed records of usage required);
3. History of chronic pain or substance abuse, such as opioids;
4. Diagnosed mental disorders with psychotropic medication use for over 3 months prior to the visit, or history of psychotropic or hormonal medication use for over 3 months;
5. Individuals at risk of self-harm or suicide, as assessed by a psychiatrist, or those requiring psychosomatic intervention;
6. History of allergy to psychiatric medications (e.g., fluoxetine), or contraindications to fluoxetine such as liver/kidney impairment or prolonged Q-T interval on ECG;
7. Pregnant or breastfeeding women;
8. Patients with benign or malignant tumors or autoimmune diseases;
9. Chronic conditions requiring long-term medication that may affect quality of life or interfere with examinations/treatment, including cardiovascular diseases, coagulation disorders or regular anticoagulant use (warfarin/heparin), liver/kidney diseases, organ failure, cognitive impairment, aphasia, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion (%) of patients who achieved an increase of ≥1 CSBM per week compared to baseline for at least 2 out of the 4 treatment weeks. | 1-4 treatment week

SECONDARY OUTCOMES:
Proportion of participants achieving an increase of ≥1 CSBM from baseline in at least 2 weeks during follow-up | Weeks 1-4 follow-up; assessed over the 4-week period
Change from baseline in weekly frequency of spontaneous bowel movements (SBM) | Baseline and each week during Weeks 1-4
Change from baseline in weekly frequency of complete spontaneous bowel movements (CSBM) | Baseline and each week during Weeks 1-4
Change from baseline in stool consistency (Bristol Stool Form Scale) for weekly SBMs | Baseline and Weeks 3-4
Change from baseline in straining score for weekly SBMs (4-point scale: 0=no difficulty, 1=mild, 2=moderate, 3=severe) | Baseline and Weeks 3-4
Change from baseline in abdominal bloating severity (5-point scale: 1=none, 2=mild, 3=moderate, 4=severe, 5=very severe) | Baseline and Weeks 3-4
Change from baseline in Patient Health Questionnaire-9 (PHQ-9) score | Baseline and Week 4
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) score | Baseline and Week 4
Change from baseline in Patient Health Questionnaire-15 (PHQ-15) somatic symptom score | Baseline and Week 4
Change from baseline in Patient Assessment of Constipation-Quality of Life (PAC-QOL) | Baseline and Week 4
Proportion of participants using polyethylene glycol (PEG) as rescue medication | During the 4-week treatment period

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact zhaozhifeng@outlook.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: For more information or to submit a request, please contact zhaozhifeng@outlook.com.
URL: https://prsinfo.clinicaltrials.gov/definitions.html